CLINICAL TRIAL: NCT02269410
Title: Metabolic Impact of Dietary Protein Supplementation in Surgical Weight Loss II (MIPS II)
Brief Title: Metabolic Impact of Dietary Protein Supplementation in Surgical Weight Loss
Acronym: MIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Blandine Laferrere, Associate professor of medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAN6105
Record Dates: First submitted 2014-10-10; First posted 2014-10-21 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Obesity
Keywords: Bariatric Surgery; Nitrogen Balance; Body composition; Protein supplementation; Satiety; Adherence
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- GBP-SPS (Active Comparator): GBP Standard PRO-S (0.8g protein/kg ideal body weigh/day)
  Interventions: Dietary Supplement: GBP-SPS
- GBP-HPS (Experimental): GBP High PRO-S (1.2g protein/ kg ideal body weight/ day)
  Interventions: Dietary Supplement: GBP-HPS
- VSG-SPS (Active Comparator): VSG Standard PRO-S (0.8g protein/kg ideal body weigh/ day)
  Interventions: Dietary Supplement: VSG-SPS
- VSG-HPS (Experimental): VSG High PRO-S (1.2g protein/ kg ideal body weight/ day)
  Interventions: Dietary Supplement: VSG-HPS

INTERVENTIONS:
Dietary Supplement: GBP-SPS — Protein powder supplementation will be given to participants to add to regular foods during the dietary intervention phase until reach protein objectives based on randomization and during 12 weeks after Bariatric Surgery.
  Arms: GBP-SPS
Dietary Supplement: GBP-HPS — Protein powder supplementation will be given to participants to add to regular foods during the dietary intervention phase until reach protein objectives based on randomization and during 12 weeks after Bariatric Surgery.
  Arms: GBP-HPS
Dietary Supplement: VSG-SPS — Protein powder supplementation will be given to participants to add to regular foods during the dietary intervention phase until reach protein objectives based on randomization and during 12 weeks after Bariatric Surgery.
  Arms: VSG-SPS
Dietary Supplement: VSG-HPS — Protein powder supplementation will be given to participants to add to regular foods during the dietary intervention phase until reach protein objectives based on randomization and during 12 weeks after Bariatric Surgery.
  Arms: VSG-HPS

SUMMARY:
The obesity epidemic has grown rapidly in the United States, and is associated with increased morbidity and mortality rates. Bariatric surgery (BS) has emerged as the most effective treatment for severe obesity. Surgical weight loss (WL) is very significant (~40-50kg) during the first 6-12 months after surgery. The adequate amount of dietary protein during the active period of surgical weight loss is not known. Dietary protein affects body weight regulation: satiety, thermogenesis, energy efficiency and body composition. During diet-induced energy-restriction, sustaining protein intake (PI) at the level of requirement (0.8g /kg ideal body weight (IBW)/ day) appears to preserve fat free mass (FFM) during active WL. PI above requirements (1.2g protein/Kg IBW/ day) results in favorable body composition changes, with greater decrease in fat mass and preservation of FFM, but without effecting WL. Dietary PI 0.8g/day has been associated with greater satiety and increased energy expenditure (EE) during calorie restriction. In this randomized prospective study, the investigators will evaluate the effect of PI on nitrogen balance, body composition, EE and satiety in 40 women undergoing either Gastric Bypass or Vertical Sleeve Gastrectomy, assigned to high protein supplementation (PRO-S), high PRO-S (1.2g /kg IBW/day) or standard- based current guidelines -PRO-S (0.8g /kg IBW/day). PRO-S will be supplied for 3 months after surgery. Outcome measures including nitrogen balance, body composition changes and satiety will be assessed at pre-surgery, and at 3, 6 and 12 months post-surgery. These results will help provide evidence-based data on safe and optimal levels of protein supplementation after BS

DETAILED DESCRIPTION:
The goal of this proposal is to study the effect of dietary protein supplementation (PRO-S) during surgical weight loss, on nitrogen balance, energy expenditure, body composition of weight loss, and satiety. The overall goal is to provide evidence-based data on optimal levels of protein supplementation after surgical weight loss by gastric bypass (GBP), a restrictive and malabsorptive procedure, or by vertical sleeve gastrectomy (VSG), a purely restrictive procedure.

We propose a prospective randomized controlled trial (RCT), in which, patients undergoing either GBP or VSG will be allocated to standard PRO-S recommendation ("standard care" according to the American Society for Metabolic and Bariatric Surgery Guidelines) or high supplementation. We will compare 4 groups of subjects:

* Group 1: GBP Standard PRO-S (0.8g protein/kg ideal body weight (IBW)/day
* Group 2: GBP High PRO-S (1.2g protein/ kg ideal body weight (IBW)/ day)
* Group 3: VSG Standard PRO-S (0.8g protein/kg ideal body weight (IBW)/day
* Group 4: VSG High PRO-S (1.2g protein/ kg ideal body weight (IBW)/ day)

AIM#1: Measure total body nitrogen balance (NB) to assess adequacy of levels of protein intake and protein absorption.

AIM#2: Measure the effect PRO-S on lean body mass (LBM), and resting energy expenditure (REE).

AIM#3: Measure the effect of PRO-S on satiety. Hypothesis 3.1: Patients in the High PRO-S group will experience higher levels of perceived satiety compared with patients in the standard PRO-S group.

AIM #4: Study adherence to protein supplementation. Hypothesis : Adherence will be greater in the Standard PRO-S group.

Background and Significance The obesity epidemic has grown rapidly in the United States, and is associated with increased morbidity and mortality rates. Although preventive measures are needed to solve the obesity epidemic in the long-term, bariatric surgery has become a popular and effective treatment of severe obesity. Obesity and its co-morbidities, including type 2 diabetes (T2DM), have a high health care cost2. The cost is even greater for severe obesity (BMI≥40 kg/m2).

Protein (PRO) malnutrition after bariatric surgery (BS) Bariatric surgery (BS) has emerged as the most effective treatment for severe obesity. Gastric bypass surgery (GBP) results in large weight loss with normalization of metabolic functions, including T2DM remission in ~60-80% of cases. Weight loss is very significant (~40-50kg). The rate of weight loss is rapid during the first year after surgery. Surgical weight loss can be associated with vitamin, mineral, and protein deficiencies. PRO malnutrition, remains the most severe nutritional complication associated with malabsorptive surgical procedures. The prevalence of protein malnutrition after malabsorptive BS procedures varies between 3 to 18% and is associated with the length of the bypassed segment. The US recommended dietary allowance (RDA) for protein is ~50 g/d for healthy normal weight adults. Experts and clinicians recommend ~70 g/d of protein during low-calorie diets or 60 g/day (standard) and 120 g/day (high) in the earlier months after BS. However, there is little evidence-based data to support these recommendations. In spite of the absence of level 1 data on types and amount of protein recommendations, the American Society for Metabolic Surgery and BS's website has 14 links for commercial nutrition supplements14. In this study, we aim to study protein absorption and adequacy of protein intake by nitrogen balance in patients following standard and high PRO-S following BS.

Effects of dietary proteins Dietary PRO-S and amino acids (AA) are important modulators of body weight by affecting various determinants of body weight regulation: satiety, thermogenesis, energy efficiency and body composition. During energy restriction, sustaining protein intake at the level of requirement (0.8g protein/kg ideal body weight (IBW)/ day) appears to be sufficient to induce body weight loss while preserving fat free mass (FFM). Protein intake above requirements (1.2g protein/Kg IBW/ day) results in a greater decrease in fat mass and preservation of FFM, but has no effect on body weight loss.

Nitrogen balance (NB) study The NB method is classically used to determine adequate protein intakes and to measure whole body protein balance in response to nutritional interventions. Prolonged negative nitrogen balance should not be sustained for long periods due its negative impact on overall health.

Risk of decreased lean body mass (LBM) and resting energy expenditure (REE) with surgical weight loss BS results in large weight losses (30-50kg), with both fat mass (FML) and LBM losses. Our previous observational studies aiming to evaluate the relationship between protein intake and loss of LBM following BS have shown that protein intake > 60g/ day is associated with better maintenance of LBM after BS. LBM is the main determinant of REE, explaining 75% of the REE variance with REE being the largest component of 24-h energy expenditure (EE). Reduced EE may trigger weight regain in this population. High PRO-S diets may also benefit this population by increasing EE while preventing LBM loss. Increased EE from dietary protein is attributed to an enhanced thermic effect (23-30%) compared to carbohydrates (5-10%) or lipids (2-3%).

Dietary protein intake and satiety High-protein intake increases satiety despite energy restriction. Proposed mechanisms are as follows: a ketogenic state, relatively elevated plasma amino acid (AA) levels, and anorexigenic hormone concentrations feedback on the central nervous system to prolong the duration before one feels hunger for the next meal (satiety) such as, Peptide YY, Glucagon-Like Peptide -1 and cholecystokinin produced in response to peripheral and central detection of amino acid, and decreased levels of the orexigenic hormone ghrelin.

Protein supplementation and adherence Low protein intake after BS has been reported. PRO-S has always been recommended after BS but its feasibility has not been well addressed in any RCT. We will study adherence to PRO-S. Increasing adherence with dietary recommendation is challenging, but may represent a key strategy to improve the clinical nutritional treatment and outcomes after BS.

ELIGIBILITY:
Inclusion Criteria:

1. Women scheduled to undergo either GBP or VSG.
2. Ethnicity/gender: People of all race/ethnicity are eligible to participate, so that the study will reflect a diverse population.
3. Non diabetic or diet controlled diabetic with no medication

Exclusion Criteria:

1. Individuals who have a clinical history strongly suggestive of type 1 diabetes mellitus or T2DM will be excluded.
2. Nitrogen retention disease such as renal or hepatic disease.
3. Known malabsorption syndrome.
4. Any other condition which, in the opinion of the investigators, may make the candidate unsuitable for participation in this study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in Nitrogen balance (NB) | Change from baseline of NB at 3 months after surgery
  During inpatient stay. Nitrogen intake and output will be accurately monitored
Change in Nitrogen balance (NB) | Change form 3 month to 12 months
  During inpatient stay. Nitrogen intake and output will be accurately monitored
Change in Nitrogen Balance | Change from baselina to 12 months
  During inpatient stay. Nitrogen intake and output will be accurately monitored

SECONDARY OUTCOMES:
Composite outcome measure consisting of Lean body mass (LBM), and resting energy expenditure (REE). | 0, 3 and 12 months after surgery
  LBM (Kg) will be analyzed by Bod Pod and Total Body Water technique REE will be determined by indirect calorimetry
Satiety scores | 0, 3 and 12 months
  Hormonals levels and perceived satiety scores will be evaluated
Adherence score to protein supplementation. | 0, 3 and 12 months
  Score of Adherence will be obtained

CONTACTS AND LOCATIONS:
Overall Officials: Blandine Laferrere, MD, Principal Investigator — Columbia University; Xavier Pi-Sunyer, MD, Principal Investigator — Columbia University

REFERENCES:
- [Background] Buchwald H, Estok R, Fahrbach K, Banel D, Jensen MD, Pories WJ, Bantle JP, Sledge I. Weight and type 2 diabetes after bariatric surgery: systematic review and meta-analysis. Am J Med. 2009 Mar;122(3):248-256.e5. doi: 10.1016/j.amjmed.2008.09.041. PMID 19272486
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Shah M, Simha V, Garg A. Review: long-term impact of bariatric surgery on body weight, comorbidities, and nutritional status. J Clin Endocrinol Metab. 2006 Nov;91(11):4223-31. doi: 10.1210/jc.2006-0557. Epub 2006 Sep 5. PMID 16954156
- [Background] Byrne TK. Complications of surgery for obesity. Surg Clin North Am. 2001 Oct;81(5):1181-93, vii-viii. doi: 10.1016/s0039-6109(05)70190-0. PMID 11589251
- [Background] Stocker DJ. Management of the bariatric surgery patient. Endocrinol Metab Clin North Am. 2003 Jun;32(2):437-57. doi: 10.1016/s0889-8529(03)00002-1. PMID 12800540
- [Background] Skroubis G, Sakellaropoulos G, Pouggouras K, Mead N, Nikiforidis G, Kalfarentzos F. Comparison of nutritional deficiencies after Roux-en-Y gastric bypass and after biliopancreatic diversion with Roux-en-Y gastric bypass. Obes Surg. 2002 Aug;12(4):551-8. doi: 10.1381/096089202762252334. PMID 12194550
- [Background] Brolin RE, Kenler HA, Gorman JH, Cody RP. Long-limb gastric bypass in the superobese. A prospective randomized study. Ann Surg. 1992 Apr;215(4):387-95. doi: 10.1097/00000658-199204000-00014. PMID 1558421
- [Background] Dodell GB, Albu JB, Attia L, McGinty J, Pi-Sunyer FX, Laferrere B. The bariatric surgery patient: lost to follow-up; from morbid obesity to severe malnutrition. Endocr Pract. 2012 Mar-Apr;18(2):e21-5. doi: 10.4158/EP11200.CR. PMID 22138075
- [Background] Kushner R. Managing the obese patient after bariatric surgery: a case report of severe malnutrition and review of the literature. JPEN J Parenter Enteral Nutr. 2000 Mar-Apr;24(2):126-32. doi: 10.1177/0148607100024002126. PMID 10772194
- [Background] Mechanick JI, Youdim A, Jones DB, Timothy Garvey W, Hurley DL, Molly McMahon M, Heinberg LJ, Kushner R, Adams TD, Shikora S, Dixon JB, Brethauer S. Clinical practice guidelines for the perioperative nutritional, metabolic, and nonsurgical support of the bariatric surgery patient--2013 update: cosponsored by American Association of Clinical Endocrinologists, the Obesity Society, and American Society for Metabolic & Bariatric Surgery. Surg Obes Relat Dis. 2013 Mar-Apr;9(2):159-91. doi: 10.1016/j.soard.2012.12.010. Epub 2013 Jan 19. PMID 23537696
- [Background] Keller U. Dietary proteins in obesity and in diabetes. Int J Vitam Nutr Res. 2011 Mar;81(2-3):125-33. doi: 10.1024/0300-9831/a000059. PMID 22139563
- [Background] Soenen S, Martens EA, Hochstenbach-Waelen A, Lemmens SG, Westerterp-Plantenga MS. Normal protein intake is required for body weight loss and weight maintenance, and elevated protein intake for additional preservation of resting energy expenditure and fat free mass. J Nutr. 2013 May;143(5):591-6. doi: 10.3945/jn.112.167593. Epub 2013 Feb 27. PMID 23446962
- [Background] Laferrere B, Reilly D, Arias S, Swerdlow N, Gorroochurn P, Bawa B, Bose M, Teixeira J, Stevens RD, Wenner BR, Bain JR, Muehlbauer MJ, Haqq A, Lien L, Shah SH, Svetkey LP, Newgard CB. Differential metabolic impact of gastric bypass surgery versus dietary intervention in obese diabetic subjects despite identical weight loss. Sci Transl Med. 2011 Apr 27;3(80):80re2. doi: 10.1126/scitranslmed.3002043. PMID 21525399
- [Background] Energy and protein requirements: report of a joint FAO-WHO ad hoc expert committee. Rome, 22 March - 2 April 1971. World Health Organ Tech Rep Ser. 1973;522:1-118. No abstract available. PMID 4634202
- [Background] Energy and protein requirements. Report of a joint FAO/WHO/UNU Expert Consultation. World Health Organ Tech Rep Ser. 1985;724:1-206. No abstract available. PMID 3937340
- [Background] Moize V, Andreu A, Rodriguez L, Flores L, Ibarzabal A, Lacy A, Jimenez A, Vidal J. Protein intake and lean tissue mass retention following bariatric surgery. Clin Nutr. 2013 Aug;32(4):550-5. doi: 10.1016/j.clnu.2012.11.007. Epub 2012 Nov 14. PMID 23200926
- [Background] Cunningham JJ. Body composition as a determinant of energy expenditure: a synthetic review and a proposed general prediction equation. Am J Clin Nutr. 1991 Dec;54(6):963-9. doi: 10.1093/ajcn/54.6.963. PMID 1957828
- [Background] Nair KS, Halliday D, Garrow JS. Thermic response to isoenergetic protein, carbohydrate or fat meals in lean and obese subjects. Clin Sci (Lond). 1983 Sep;65(3):307-12. doi: 10.1042/cs0650307. PMID 6347500
- [Background] Blom WA, Lluch A, Stafleu A, Vinoy S, Holst JJ, Schaafsma G, Hendriks HF. Effect of a high-protein breakfast on the postprandial ghrelin response. Am J Clin Nutr. 2006 Feb;83(2):211-20. doi: 10.1093/ajcn/83.2.211. PMID 16469977
- [Background] Martens EA, Westerterp-Plantenga MS. Protein diets, body weight loss and weight maintenance. Curr Opin Clin Nutr Metab Care. 2014 Jan;17(1):75-9. doi: 10.1097/MCO.0000000000000006. PMID 24310056
- [Background] Leidy HJ, Carnell NS, Mattes RD, Campbell WW. Higher protein intake preserves lean mass and satiety with weight loss in pre-obese and obese women. Obesity (Silver Spring). 2007 Feb;15(2):421-9. doi: 10.1038/oby.2007.531. PMID 17299116
- [Background] Faria SL, Faria OP, Lopes TC, Galvao MV, de Oliveira Kelly E, Ito MK. Relation between carbohydrate intake and weight loss after bariatric surgery. Obes Surg. 2009 Jun;19(6):708-16. doi: 10.1007/s11695-008-9583-y. Epub 2008 Jul 10. PMID 18618210
- [Background] Moize V, Andreu A, Flores L, Torres F, Ibarzabal A, Delgado S, Lacy A, Rodriguez L, Vidal J. Long-term dietary intake and nutritional deficiencies following sleeve gastrectomy or Roux-En-Y gastric bypass in a mediterranean population. J Acad Nutr Diet. 2013 Mar;113(3):400-410. doi: 10.1016/j.jand.2012.11.013. PMID 23438491
- [Background] Wang TJ, Larson MG, Vasan RS, Cheng S, Rhee EP, McCabe E, Lewis GD, Fox CS, Jacques PF, Fernandez C, O'Donnell CJ, Carr SA, Mootha VK, Florez JC, Souza A, Melander O, Clish CB, Gerszten RE. Metabolite profiles and the risk of developing diabetes. Nat Med. 2011 Apr;17(4):448-53. doi: 10.1038/nm.2307. Epub 2011 Mar 20. PMID 21423183
- [Background] Trumbo P, Schlicker S, Yates AA, Poos M; Food and Nutrition Board of the Institute of Medicine, The National Academies. Dietary reference intakes for energy, carbohydrate, fiber, fat, fatty acids, cholesterol, protein and amino acids. J Am Diet Assoc. 2002 Nov;102(11):1621-30. doi: 10.1016/s0002-8223(02)90346-9. No abstract available. PMID 12449285
- [Background] Levitt DG, Beckman LM, Mager JR, Valentine B, Sibley SD, Beckman TR, Kellogg TA, Ikramuddin S, Earthman CP. Comparison of DXA and water measurements of body fat following gastric bypass surgery and a physiological model of body water, fat, and muscle composition. J Appl Physiol (1985). 2010 Sep;109(3):786-95. doi: 10.1152/japplphysiol.00278.2010. Epub 2010 Jun 17. PMID 20558754
- [Background] Widen EM, Strain G, King WC, Yu W, Lin S, Goodpaster B, Thornton J, Courcoulas A, Pomp A, Gallagher D. Validity of bioelectrical impedance analysis for measuring changes in body water and percent fat after bariatric surgery. Obes Surg. 2014 Jun;24(6):847-54. doi: 10.1007/s11695-014-1182-5. PMID 24464517
- [Background] Rosenbaum M, Ravussin E, Matthews DE, Gilker C, Ferraro R, Heymsfield SB, Hirsch J, Leibel RL. A comparative study of different means of assessing long-term energy expenditure in humans. Am J Physiol. 1996 Mar;270(3 Pt 2):R496-504. doi: 10.1152/ajpregu.1996.270.3.R496. PMID 8780213
- [Background] Cardello AV, Schutz HG, Lesher LL, Merrill E. Development and testing of a labeled magnitude scale of perceived satiety. Appetite. 2005 Feb;44(1):1-13. doi: 10.1016/j.appet.2004.05.007. Epub 2004 Nov 13. PMID 15604029
- [Derived] Moize V, Pi-Sunyer X, Vidal J, Miner P, Boirie Y, Laferrere B. Effect on Nitrogen Balance, Thermogenesis, Body Composition, Satiety, and Circulating Branched Chain Amino Acid Levels up to One Year after Surgery: Protocol of a Randomized Controlled Trial on Dietary Protein During Surgical Weight Loss. JMIR Res Protoc. 2016 Nov 28;5(4):e220. doi: 10.2196/resprot.6438. PMID 27895003
- See also: Obesity Update 2012 — http://www.oecd.org/health/49716427.pdf
- See also: Unit States Department of agriculture — http://www.nal.usda.gov/fnic